CLINICAL TRIAL: NCT00422539
Title: Evaluation of Tri Chloro Acetic Acid (TCA) Effect on Atrophic Varicella Scars
Brief Title: Efficacy of TCA Effect on Varicella Atrophic Scars
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRC-BBA-1385-6-1
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Atrophic Varicella Scar
Keywords: trichloroacetic acid; varicella scar
MeSH Terms: interventions — Trichloroacetic Acid

INTERVENTIONS:
Drug: 70% trichloroacetic acid

SUMMARY:
This study aims to determine the efficacy of 70% trichloroacetic acid on atrophic scars of varicella

DETAILED DESCRIPTION:
high concentration trichloroacetic acid peeling has been shown to be effective in treating and flattening the atrophic acne scars. According to the lack of an effective and low cost therapy for removing these relative common and nuisance lesions; We aimed to answer that whether we could achieve the same results from 70% TCA on atrophic varicella scars.

ELIGIBILITY:
Inclusion Criteria:

* Atrophic varicella scar on face

Exclusion Criteria:

* Active varicella infection
* Active Herpetic infection
* Previous history of keloid formation

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2006-03

PRIMARY OUTCOMES:
Objective Clearance(before and after photographies were taken)

SECONDARY OUTCOMES:
Subjective Clearance(according to the patients satisfaction)
Adverse effects(assessed by clinician as erythema, pigmentary changes, scaring)

CONTACTS AND LOCATIONS:
Overall Officials: Parviz Toossi, M.D., Study Chair — Skin Research Center of Shaheed Beheshti medical University; Behrooz Barikbin, M.D., Principal Investigator — Skin Research Center of Shaheed Beheshti Medical Universty
Locations (1):
- Skin Research Center, Shohada-e Tajrish Hospital, shaheed Beheshti Medical University, Tehran, Tehran Province, Iran